CLINICAL TRIAL: NCT06223425
Title: Effectiveness of Virtual Reality Situation-Based Flipped Learning and Gamification on Nursing Students' Learning Attitudes, Problem-solving Abilities, and Empathetic Abilities
Brief Title: Virtual Reality Situation-Based Flipped Learning
Acronym: VRFlipped
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00013623
Record Dates: First submitted 2024-01-02; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Educational Problems; Problem;Learning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality Situation-Based Flipped Learning (Experimental): students exposed to virtual reality Situation-Based Flipped Learning
  Interventions: Behavioral: virtual reality Situation-Based Flipped Learning
- traditional teaching strategies (No Intervention): Students exposed to traditional Learning

INTERVENTIONS:
Behavioral: virtual reality Situation-Based Flipped Learning — Situation-Based Flipped Learning, and Gamification have gained attention as promising tools to engage nursing students and promote a deeper understanding of complex concepts. This study aims to investigate the effectiveness of combining these strategies in a virtual reality Situation-Based Flipped Learning environment with elements of Gamification on nursing students' learning attitudes, problem-solving abilities, and empathetic skills.
  Arms: virtual reality Situation-Based Flipped Learning

SUMMARY:
The integration of innovative educational approaches in nursing education has become increasingly crucial for enhancing learning outcomes. Among these approaches, virtual reality (VR)

DETAILED DESCRIPTION:
Situation-Based Flipped Learning, and Gamification have gained attention as promising tools to engage nursing students and promote a deeper understanding of complex concepts. This study aims to investigate the effectiveness of combining these strategies in a virtual reality Situation-Based Flipped Learning environment with elements of Gamification on nursing students' learning attitudes, problem-solving abilities, and empathetic skills. By leveraging these technologies, educators seek to create an immersive and interactive learning experience that not only aligns with the demands of modern education but also addresses the unique challenges faced by nursing students in developing critical competencies. This research explores the potential impact of this integrated approach on nursing education, contributing valuable insights to the ongoing efforts to optimize teaching methodologies for future healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate

Exclusion Criteria:

* First-year academic students

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
virtual reality Situation-Based Flipped Learning | two months
  Students who were exposed to virtual reality Situation-Based Flipped Learning and Gamification exhibited a higher level of Problem-Solving Ability measured by the Problem-Solving Ability scale (a higher score of more than 90) than those in traditional learning strategies
virtual reality Based Gamification | two months
  students who were exposed to virtual reality Situation-Based Flipped Learning and Gamification exhibited a higher level of empathic understanding level measured by the Empathetic ability scale ( a higher score of more than15) than those in traditional learning strategies

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H atta, Principal Investigator — Faculty of nursing, Alexandria university, Egypt
Locations (1):
- Alexandria university, Alexandria, Alexandria Governorate, Egypt

DOCUMENTS (1):
  • Study Protocol (2024-01-10): https://cdn.clinicaltrials.gov/large-docs/25/NCT06223425/Prot_000.pdf